CLINICAL TRIAL: NCT06558877
Title: Effect of a Pharmacist-led Multifaceted Intervention on Treatment Outcomes in Hypertensive Patients: a Cluster Randomised Clinical Trial
Brief Title: Effect of a Pharmacist-led Multifaceted Intervention on Treatment Outcomes in Hypertensive Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Sichuan Academy of Medical Sciences (Other); Zhejiang University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); The People's Hospital of Shaanxi Province (Unknown); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Tang-Du Hospital (Other); LanZhou University (Other)
Responsible Party: Principal Investigator, Wang Jingwen, Director of Pharmacy Department, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KY20242276
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental)
  Interventions: Behavioral: pharmacist-led multifaceted intervention
- control group (Other)
  Interventions: Behavioral: conventional health education

INTERVENTIONS:
Behavioral: pharmacist-led multifaceted intervention — Based on the blood pressure management model of pharmacist-led multifaceted intervention, clinical pharmacists who have received unified training provide pharmaceutical intervention and lifestyle guidance to subjects in the intervention group according to standard protocol.
  Pharmaceutical interventions include health education, medication adherence (medication consultation, medication reminder), medication reorganization, and rational use of medication. At the same time, clinical pharmacists supervise the subjects to change their lifestyle (including reasonable diet, quitting smoking and drinking, moderate exercise, weight control and ensuring sleep, etc.), and guide the subjects to conduct home blood pressure monitoring.
  Arms: intervention group
Behavioral: conventional health education — The subjects receive conventional hypertension health education, standard blood pressure measurement training and regular follow-up in the control group.
  Arms: control group

SUMMARY:
The objective of this cluster randomized controlled trial is to evaluate the effectiveness of a pharmacist-led multifaceted intensive blood pressure intervention on poorly controlled hypertensive patients in phase 1 (1 month, 3 months, 6 months, 12 months) and phase 2 (24 months) post randomization.

DETAILED DESCRIPTION:
This cluster randomized trial is conducted in eight tertiary hospitals of China, and we planned to enroll 100 participants at each hospital. The eight hospitals will be randomly divided into an intervention group or a control group in a 1:1 ratio. A total of 800 patients with poorly controlled blood pressure aged 18-80 years will be recruited into the study. The pharmacist-led multifaceted intervention is comprised of all the following five components: 1) Health education: lectures on hypertension related knowledge, the potential risks of hypertension, and guidance on healthy lifestyle, etc; 2) home blood pressure telemonitoring; 3) Medication consultation: including the usage, dosage, precautions and adverse reactions of hypertension drugs; 4) Medication reminders: remind subjects to take medication on time by Wechat or Messages; 5) Formulation of individualized medication regimen: efficacy evaluation and drug realignment. However, the control group received routine hypertension health education, standardized blood pressure measurement and regular follow-up.

The primary outcome is to assess the change in blood pressure control rate, time in target range (TTR), adherence to antihypertensive medication rate, and cardiovascular disease (CVDs) between the intervention group and the control group from baseline to follow-up at 1 month, 3 months, 6 months, 12 and 24 months post randomization. The secondary outcome is to assess the change in the mean systolic and diastolic pressures, and the medication appropriateness measured by the medication appropriateness index (MAI) between the two groups in phase 1 and 2. Meanwhile, the BMI, alcohol use and smoking will be also assessed in phase 1, and the incidence of hypertension-related adverse events will be assessed in phase 2.

ELIGIBILITY:
Inclusion Criteria (subjects must meet all of the following criteria to be included):

* 1) age 18-80 years;
* 2) patients with hypertension (diagnostic criteria: defined as systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg according to the "Guidelines for the prevention and treatment of hypertension in China in 2023", based on the blood pressure measurement of three times on different days), who are currently taking anti-hypertensive medication and are judged by the research physician to have poor blood pressure control;
* 3) able to use smartphones and WeChat proficiently, and can communicate and upload pictures proficiently;
* 4) able to take care of yourself and communicate normally, and willing to cooperate with the research physician to complete the study and follow-up;
* 5) permanent residents of the city where the center is located;
* 6) voluntarily participate and sign the informed consent form

Exclusion Criteria(subjects will be excluded if they meet any of the following criteria):

* 1) patients with advanced disease (such as patients undergoing dialysis or liver failure), or with a life expectancy of less than 2 years as determined by the research physician;
* 2) combined with psychiatric disease, cognitive impairment, communication disorder, or inability to cooperate with the researchers;
* 3) combined with cerebrovascular disease, stroke, severe liver and kidney dysfunction, severe heart failure, cancer and history of organ transplantation, etc.;
* 4) patients who are pregnant, breastfeeding, or planning to conceive in the next 2 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure control rate | baseline, 1 month, 3 months, 6 months, 12 months and 24 months after baseline
  The proportion of participants with controlled blood pressure
Time in target range (TTR) | baseline, 1 month, 3 months, 6 months, 12 months and 24 months after baseline
  TTR is the proportion of time that a subject's blood pressure value is within the specified target blood pressure range, which reflects the average blood pressure (BP) value and the degree of blood pressure variability during long-term follow-up.
Medication Adherence | baseline, 1 month, 3 months, 6 months and 12 months after baseline
  The Morisky Medication Adherence Scale is used for evaluating the medication adherence. Compare the change in medication adherence between the intervention group and the control group. The 8 items version of the Morisky will be used, and Morisky score will range from 0 to 8. Higher scores indicate better medication adherence.
Cardiovascular events and all-cause death | baseline and 24 months after baseline
  Record cardiovascular events and all-cause death

SECONDARY OUTCOMES:
Mean systolic and diastolic pressure changes | baseline, 1 month, 3 months, 6 months, 12 months and 24 months after baseline
  Mean systolic and diastolic pressure changes of participants
Medication Appropriateness Index | baseline, 1 month, 3 months, 6 months, 12 months and 24 months after baseline
  Medication Appropriateness Index (MAI), assessed at baseline as well as at the 1, 3, 6 and 12 months follow-ups for each patient. The 10 items version of the MAI will be used, and the MAI score for each medication will range from 0 to 17. Higher scores indicate worse medication appropriateness.
Body Mass Index (BMI) | baseline, 1 month, 3 months, 6 months and 12 months after baseline
  Measure height and weight of subjects, and calculate BMI. Compare the change in BMI of subjects between the intervention group and the control group.
Alcohol consumption | baseline, 1 month, 3 months, 6 months and 12 months after baseline
  Record alcohol consumption by Alcohol Use Disorders Identification Test (AUDIT). The 10 items version of the AUDIT will be used, and AUDIT score will range from 0 to 40. Higher scores indicate greater alcohol dependence.
Nicotine consumption | baseline, 1 month, 3 months, 6 months and 12 months after baseline
  The smoking behavior, measured by fagerstrom test of nicotine dependence (FTND) scale in smoking patients from baseline to follow-up at 1, 3, 6 and 12 months. The 6 items version of the FTND will be used, and the FTND score will range from 0 to 10. Higher scores indicate greater nicotine dependence.
Medication Adherence | baseline and 24 months after baseline
  The Morisky Medication Adherence Scale is used for evaluating the medication adherence. Compare the change in medication adherence between the intervention group and the control group. The 8 items version of the Morisky will be used, and Morisky score will range from 0 to 8. Higher scores indicate better medication adherence.
Patients' medical costs | baseline, 1 month, 3 months, 6 months and 12 months after baseline
  Comparison of the direct medical costs between the intervention and control groups during one year.
Hypertension-related adverse events rate | baseline and 24 months after baseline
  Proportion of participants with hypertension-related adverse events (include hypotension, syncope, traumatic falls, bradycardia, electrolyte abnormalities, or acute kidney injury)

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided